CLINICAL TRIAL: NCT04737889
Title: A Single Arm, Multi-center, Phase II Clinical Trial of Rituximab, Lenalidomide Combined With High-dose Methotrexate and Temozolomide (RL-MT) in the First-line Treatment for Patients With Primary Central Nervous System Lymphoma
Brief Title: Rituximab, Lenalidomide Combined With Methotrexate and Temozolomide For Primary Central Nervous System Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhihua Yao, PhD, Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYYNHL04
Record Dates: First submitted 2021-01-30; First posted 2021-02-04 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Primary Central Nervous System Lymphoma; RL-MT
MeSH Terms: interventions — Rituximab; Lenalidomide; Methotrexate; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RL-MT (Experimental): Induction Chemotherapy: Rituximab, 375mg/m2, Intravenous administration on day 0, Lenalidomide, 25mg oral administration on day 1 to 10, combined with regimen: Methotrexate, 3mg/m2, Intravenous administration (pumping for 3h) on day 1 of each 3-week cycle, Temozolomide, 150mg/m2/d oral administration on day 1 to 10.
  Consolidation Treatment: Autologous hematopoietic stem cell transplantation or reduced whole brain radiotherapy after high-dose chemotherapy.
  Maintenance Treatment: Lenalidomide, 10mg oral administration on day 1 to 21 of each 4-week cycle for 12 months.
  Interventions: Drug: Rituximab; Drug: Lenalidomide; Drug: Methotrexate; Drug: Temozolomide

INTERVENTIONS:
Drug: Rituximab — Induction Chemotherapy: 375mg/m2, Intravenous administration on day 0 of each 3-week cycle until disease progression/stable disease or unacceptable toxicity develops, up to 6 cycles.
  Other Names: RiTUXimab Injection
Drug: Lenalidomide — Induction Chemotherapy: 25mg, oral administration on day 1 to 10 of each 3-week cycle until disease progression/stable disease or unacceptable toxicity develops, up to 6 cycles.
  Maintenance Treatment: 10mg oral administration on day 1 to 21 repeated every 4 weeks until disease progression or unacceptable toxicity develops, up to 12 cycles.
  Other Names: Lenalidomide capsule
Drug: Methotrexate — Induction Chemotherapy: 3mg/m2, Intravenous administration (pumping for 3h) on day 1 of each 3-week cycle until disease progression/stable disease or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Methotrexate Injectable Solution
Drug: Temozolomide — Induction Chemotherapy: 150mg/m2/d oral administration on day 1 to 10 of each 3-week cycle until disease progression/stable disease or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Temozolomide capsule

SUMMARY:
This is a prospective single arm, multi-center, phase II clinical trial to observe the efficacy and safety of Rituximab, Lenalidomide combined with high-dose Methotrexate and Temozolomide (RL-MT) in the first-line treatment for patients with primary central nervous system lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 70 years old (including 18 and 70)
2. Diagnosed as primary central nervous system lymphoma (limited to the brain, spinal cord, meninges and eyeballs, without involvement of other parts)
3. Having not received anti-tumor therapy before enrollment (except for tumor resection and biopsy and the use of glucocorticoids to reduce central nervous system symptoms)
4. Having at least one measurable lesions
5. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-2 ( ECOG 3 due to tumors can be included after being fully assessed by the investigator)
6. Life expectancy no less than 1 month
7. enough main organ function
8. Pregnancy test within 7 days must be negative for women of childbearing period, and appropriate measures should be taken for contraception for women in childbearing period during the study and six months after this study
9. Agreeing to sign the written informed consents

Exclusion Criteria:

1. Diagnosed as secondary central nervous system lymphoma
2. Diagnosed as CD20 negative large B cell primary central nervous system lymphoma
3. Active malignant tumor need be treated at the same time
4. Other malignant tumor history
5. Serious surgery and trauma less than two weeks
6. Patients with active tuberculosis
7. Systemic therapy for serious acute/chronic infection
8. Congestive heart failure, uncontrolled coronary heart disease, arrhythmia and heart infarction less than 6 months
9. HIV-positive, AIDS patients and untreated active hepatitis
10. Patients with a history of deep vein thrombosis or pulmonary embolism less than 12 months
11. Patients with a history of mental illness or drug abuse
12. Poor compliance during the trial and/or follow-up phase
13. Allergies or people who are known to be allergic to any active ingredients, excipients, mouse-derived products or heterologous protein contained in this trial
14. Researchers determine unsuited to participate in this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-01-13 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | from the day of the first cycle of treatment to the date of confirmed progressive disease or death, whichever occurs first, up to 2 years after last patient's enrollment (each cycle is 21 days)
  the total proportion of patients with no progression from date of the first day of treatment to the date of confirmed progressive disease or death which one occurs first

SECONDARY OUTCOMES:
objective response rate | every 6 weeks from the day of the first cycle of induction chemotherapy treatment and every 8 weeks from the day of the first cycle of maintenance treatment to 18 months after last patient's enrollment (each cycle is 21 days)
  the total proportion of patients with complete response (CR) and partial response (PR)
overall survival | from date of the first cycle of treatment to the date of death from any cause, assessed up to 5 years (each cycle is 21 days)
  from date of first day of treatment to the date of death by any cause
incidence and relationship with study drugs of grade 3-4 adverse events | from the date of the first cycle of treatment to 18 months after last patient's enrollment (each cycle is 21 days)
  the incidence and relationship with study drugs of grade 3 or 4 adverse events (based on NCI CTC-AE v4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Yao, M.D. Ph.D, Study Director — Henan Cancer Hospital; Yanyan Liu, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China